CLINICAL TRIAL: NCT04815122
Title: Correlation Between the Presence of COMT Val158Met Polymorphism and Dopaminergic Transporter Density (DAT) in Obese Young Women
Brief Title: Correlation Between COMT Val158Met Polymorphism and Dopaminergic Transporter Density (DAT) in Obese Women
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Vivian Marques Miguel Suen, Professor of Internal Medicine Department at Ribeirão Preto Medical School, University of Sao Paulo
Other Study IDs: Process HCRP 3.844.428
Record Dates: First submitted 2021-03-05; First posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Obesity
Keywords: Obesity; Genetic polymorphism; Dopamine
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Carriers of the Met allele of the COMT Val158Met polymorphism: Women with obesity carriers of the Met allele of the COMT Val158Met polymorphism
  Interventions: Radiation: SPECT TRODAT-1
- Non-carriers of the Met allele of the COMT Val158Met polymorphism: Women with obesity non-carriers of the Met allele of the COMT Val158Met polymorphism
  Interventions: Radiation: SPECT TRODAT-1

INTERVENTIONS:
Radiation: SPECT TRODAT-1 — The Single-photon Emission Tomography (SPECT) TRODAT-1 will be performed after the voluntary rest in a dark and silent room for 30 minutes, to eliminate possible influences from external stimuli; the radiopharmaceutical [99mTC] -TRODAT-1 will be injected through the venous access previously established, 4 hours after the injection of the radiopharmaceutical, the acquisition of cerebral SPECT will be performed in the two groups of obese women, with and without COMT Val158Met polymorphism. The images will be acquired on Philips BrightView XCT equipment, equipped with a double detector.

SUMMARY:
The present study aims to evaluate the correlation between the presence of COMT Val158Met polymorphism and the density of dopaminergic transporters (DAT) in young obese women.

DETAILED DESCRIPTION:
The prevalence of obesity remains increasingly alarming in Brazil and worldwide. The most widely recommended therapy for obesity is lifestyle modification, however, implementing these changes that can lead to weight loss is difficult and maintaining a long-term weight loss is even more challenging. Consequently, an academic effort is required to understand the pathophysiology and treat obesity for the establishment of new approaches to reducing food intake.

Recent evidence in the field of obesity and brain-based integration indicates a potential for designing new therapeutic interventions. Noninvasive neuromodulation of brain activity has been shown to be a technique that can help reduce food cravings and food intake and, more recently, body weight, offering a new way to treat obesity. However, recent studies have shown that this biomedical intervention could have a paradoxical effect related to COMT Val158Met polymorphism, which impacts dopamine levels in the prefrontal cortex. The potential mechanisms underlying this effect are unclear and future studies are needed to promote this clarification.

This study aims to verify the influence of the COMT Val158Met polymorphism on the density of dopaminergic transporters in the presynaptic membrane of dopaminergic neurons, exploring the 3 dopaminergic pathways: via nigroestrital, mesolimbic and mesocortical. This investigation will be carried out through the cerebral SPECT using the radiopharmaceutical 99mTecnécio-TRODAT-1 in young obese women with and without COMT Val158Met polymorphism. In baseline conditions, the investigators will compare the SPECT 99mTc-TRODAT-1 of obese women with and without the COMT Val158Met polymorphism with a database of non-obese volunteers.

Our hypothesis is that the study will facilitate understanding of the variability of the individual response of carriers and non-carriers of the Met allele of the COMT Val158Met polymorphism, affecting dopamine levels in the brain and to design, in the future, for the treatment of obesity based on the individuals' genotypic differences.

ELIGIBILITY:
Inclusion Criteria:

* Women with obesity (BMI 30-35kg/m2), with and without COMT Val158Met polymorphism.

Exclusion Criteria:

* pregnancy
* any active psychiatric or neurological condition at the time of joining the study
* any other significant medical condition

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Young women with obesity (BMI 30-35kg/m2), with and without COMT Val158Met polymorphism who participated in a previous study registered at clinicaltrials.gov (NCT02953353).
Sampling Method: Non-Probability Sample
Enrollment: 38 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Density of Dopaminergic transporters (DAT) | During the procedure
  The primary outcome is to compare the density of dopaminergic transporters (DAT) in the 3 dopaminergic pathways: via nigroestrital, mesolimbic and mesocortical in obese women with and without COMT Val158Met polymorphism.

CONTACTS AND LOCATIONS:
Overall Officials: Vivian MM Suen, MD, PhD, Principal Investigator — University of Sao Paulo; Lauro Winchert-Ana, MD, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Clinical Hospital of Ribeirão Preto Medical School, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Avsar O, Kuskucu A, Sancak S, Genc E. Are dopaminergic genotypes risk factors for eating behavior and obesity in adults? Neurosci Lett. 2017 Jul 27;654:28-32. doi: 10.1016/j.neulet.2017.06.023. Epub 2017 Jun 16. PMID 28629779
- [Background] Barnett JH, Scoriels L, Munafo MR. Meta-analysis of the cognitive effects of the catechol-O-methyltransferase gene Val158/108Met polymorphism. Biol Psychiatry. 2008 Jul 15;64(2):137-44. doi: 10.1016/j.biopsych.2008.01.005. Epub 2008 Mar 14. PMID 18339359
- [Background] Chen PS, Yang YK, Yeh TL, Lee IH, Yao WJ, Chiu NT, Lu RB. Correlation between body mass index and striatal dopamine transporter availability in healthy volunteers--a SPECT study. Neuroimage. 2008 Mar 1;40(1):275-9. doi: 10.1016/j.neuroimage.2007.11.007. Epub 2007 Nov 21. PMID 18096411
- [Background] Fassini PG, Das SK, Suen VMM, Magerowski G, Marchini JS, da Silva Junior WA, Changyu S, Alonso-Alonso M. Appetite effects of prefrontal stimulation depend on COMT Val158Met polymorphism: A randomized clinical trial. Appetite. 2019 Sep 1;140:142-150. doi: 10.1016/j.appet.2019.05.015. Epub 2019 May 13. PMID 31095973
- [Background] Fassini PG, Das SK, Magerowski G, Marchini JS, da Silva Junior WA, da Silva IR, de Souza Ribeiro Salgueiro R, Machado CD, Suen VMM, Alonso-Alonso M. Noninvasive neuromodulation of the prefrontal cortex in young women with obesity: a randomized clinical trial. Int J Obes (Lond). 2020 Jun;44(6):1279-1290. doi: 10.1038/s41366-020-0545-3. Epub 2020 Feb 19. PMID 32076105
- [Background] Fonteneau C, Redoute J, Haesebaert F, Le Bars D, Costes N, Suaud-Chagny MF, Brunelin J. Frontal Transcranial Direct Current Stimulation Induces Dopamine Release in the Ventral Striatum in Human. Cereb Cortex. 2018 Jul 1;28(7):2636-2646. doi: 10.1093/cercor/bhy093. PMID 29688276
- [Background] Horstmann A, Fenske WK, Hankir MK. Argument for a non-linear relationship between severity of human obesity and dopaminergic tone. Obes Rev. 2015 Oct;16(10):821-30. doi: 10.1111/obr.12303. Epub 2015 Jun 22. PMID 26098597
- [Background] Van Laere K, De Ceuninck L, Dom R, Van den Eynden J, Vanbilloen H, Cleynhens J, Dupont P, Bormans G, Verbruggen A, Mortelmans L. Dopamine transporter SPECT using fast kinetic ligands: 123I-FP-beta-CIT versus 99mTc-TRODAT-1. Eur J Nucl Med Mol Imaging. 2004 Aug;31(8):1119-27. doi: 10.1007/s00259-004-1480-6. Epub 2004 Apr 3. PMID 15064872
- [Background] Slifstein M, Kolachana B, Simpson EH, Tabares P, Cheng B, Duvall M, Frankle WG, Weinberger DR, Laruelle M, Abi-Dargham A. COMT genotype predicts cortical-limbic D1 receptor availability measured with [11C]NNC112 and PET. Mol Psychiatry. 2008 Aug;13(8):821-7. doi: 10.1038/mp.2008.19. Epub 2008 Mar 4. PMID 18317466
- [Background] Volkow ND, Wang GJ, Telang F, Fowler JS, Thanos PK, Logan J, Alexoff D, Ding YS, Wong C, Ma Y, Pradhan K. Low dopamine striatal D2 receptors are associated with prefrontal metabolism in obese subjects: possible contributing factors. Neuroimage. 2008 Oct 1;42(4):1537-43. doi: 10.1016/j.neuroimage.2008.06.002. Epub 2008 Jun 13. PMID 18598772
- [Background] Wang GJ, Volkow ND, Logan J, Pappas NR, Wong CT, Zhu W, Netusil N, Fowler JS. Brain dopamine and obesity. Lancet. 2001 Feb 3;357(9253):354-7. doi: 10.1016/s0140-6736(00)03643-6. PMID 11210998